CLINICAL TRIAL: NCT03309137
Title: CHG-Lock™ Device for Bacteremia Prevention in Cardiac Surgical Intensive Care Unit Patients: An Open Label Randomized Feasibility Pilot Study
Brief Title: Device for Bacteremia Prevention in Post Cardiac Surgical Intensive Care Unit Patients
Acronym: CHG-Lock™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alison Fox-Robichaud (Other)
Collaborators: Dr. Richard Whitlock (Unknown); Dr. Julian Owen (Unknown); Pamela Benoit, RN (Unknown)
Responsible Party: Sponsor-Investigator, Alison Fox-Robichaud, Professor McMaster University and Director of Medical Education at HHS, Hamilton Health Sciences Corporation
Organization: Hamilton Health Sciences Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3654
Record Dates: First submitted 2017-09-19; First posted 2017-10-13 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Infection; Heart; Surgery, Heart, Functional Disturbance as Result; Bacteremia
Keywords: Blood stream infections; Prospective; Preventative; Randomized
MeSH Terms: conditions — Infections; Bacteremia

STUDY DESIGN:
Intervention Model Description: An Open Label Randomized Feasibility Pilot Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antiseptic device (Experimental): Patients who are randomized to receive the device will receive Chlorhexidine at a dose of 0.24-0.42 mg/installation into all intravenous lines. The intervention will be administered every 24 hrs and as needed for as long as the intravenous is in place
  Interventions: Device: Chlorhexidine flush
- Routine Care (No Intervention): Patients who are randomized to routine care (no device, no intervention) will receive normal saline flush as per standard ICU care.

INTERVENTIONS:
Device: Chlorhexidine flush — 1. For patients randomized to the CHG-LockTM device, attach a attach a BD Posiflush ™ 0.9% Sodium Chloride (Na Cl) 10ml syringe and a CHG-Lock™ device for each IV line that is to be locked. Follow hospital approved protocol for flush, volumes and hand hygiene.
     After a Catheter has been locked, before re-accessing the catheter for further sampling or infusions, all fluid should be aspirated from the catheter to clear the device of CHG, Heparin and the like. This should also confirm patency of the device.
  2. Discard the syringe and device in biohazard waste.
  3. "Blue Cap" the IV as per routine practice.
  Other Names: CHG-Lock™
  Arms: Antiseptic device

SUMMARY:
Intravenous catheters are often placed in large (central) veins in critically ill patients to provide special medications or frequent blood sampling. The body reacts to the presence of foreign material by forming a biofilm on the surface within the catheter. Either due to the patients condition or to emergency access to these intravenous lines can become infected with bacteria and reside within the biofilm. When bacteria is grown from these lines it is referred to as: a central line infection. A medical device company (ICU Medical) has obtained the rights to a device that delivers a controlled amount of a cleaning material called chlorhexidine into the catheter to prevent bacterial growth when not in use. Chlorhexidine is the standard cleaning material used on patients when cleaning the skin for surgical procedures or central intravenous catheter insertion. In laboratory tests and animal studies that chlorhexidine inhibits the growth of bacteria and fungi that often cause central line infections. This study will the first assessment in patients with central lines.

DETAILED DESCRIPTION:
Randomization Randomization will be determined using an online random number generator. "www.randomize.net". The research coordinator will randomize the patients and provide bedside staff with the devices when appropriate.

Intervention

Eligible patients that have provided informed consent will be randomized to receive:

1. Steril-flow® (CHG-Lock™) device OR
2. Usual care

Test Protocol

1. For patients randomized to the CHG-LockTM device, attach a attach a BD Posiflush ™ 0.9% Sodium Chloride (Na Cl) 10ml syringe and a CHG-Lock™ device for each IV line that is to be locked. Follow hospital approved protocol for flush, volumes and hand hygiene (see appendix I, II and III).

   After a Catheter has been locked, before re-accessing the catheter for further sampling or infusions, all fluid should be aspirated from the catheter to clear the device of CHG, Heparin and the like. This should also confirm patency of the device.
2. Discard the syringe and device in biohazard waste.
3. "Blue Cap" the IV as per routine practice.

   * There is no need to use the CHG-Lock™ device for IV lines with IV solutions infusing or those attached to an IV pressure bag, to maintain IV patency.
   * If the Central Line IV is blocked, access is done by withdraw 2-3 ml discard of blood, flush with 20 mls.
   * If a line is blocked, do not force, the order must be obtained for Cathflo and administered by a certified Cathflo nurse.
   * A CHG-Lock™ device will be applied with every intravenous flush for patients in the Active (CHG-LockTM ) arm.
   * Bedside nurses will be educated on the use of the CHG-Lock™ device.
   * The device will be used for every central line and peripheral IV instillation.
   * All locking solutions must be removed prior to access. This is standard of practice.
   * Bedside nurses will be asked to document application of the device and instillation in the medication profile.
   * Pre-printed Physician Order Set will be created to ensure compliance with device use and protocol.
   * A box with devices will be placed at the bedside to ensure ease of access for nurses and that patients receive the device at every lock episode.

Duration of intervention:

* The intervention will be used while the central line or peripheral IV remains in situ.
* The intervention will be discontinued when the patient leaves the ICU or the IV is discontinued.

Measures to be taken to ensure compliance:

1. Study boxes labeled with patient name and ID at the bedside.
2. Staff education (see 3.13)
3. Daily oversight by research coordinator/Assistant

ELIGIBILITY:
Inclusion Criteria:

1. 18-100 year old adult patients admitted to the ICU;
2. Same-day admit to ICU;
3. Post-op patient with central lines in situ (PICC, multi-lumen, side arm of introducer catheters or temporary dialysis lines), AND;
4. Expected to have at least 1 central line in situ for more than 72 hrs.

Exclusion Criteria:

1. >24hrs post-admittance to ICU
2. Hopeless prognosis
3. Currently admitted with known infection or suspicion of infection (i.e. known endocarditis or other infections).
4. Chronic indwelling central venous catheters present
5. Patients with known allergies to chlorhexidine

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-19 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Compliance with the protocol | Through study completion, an average of 14 days
  The investigators will consider our study successful if we achieve compliance of than 90% use of device for locking.

SECONDARY OUTCOMES:
Bacteremia | Through study completion, an average of 14 days
  Rates of bacteremia determined by blood cultures obtained through a central line
Bacteria colonization of central line | Through study completion, an average of 14 days
  Central Line Colonization Testing will be completed when the investigators are able to obtain the discontinued central line catheters for Electron Microscopy examination

CONTACTS AND LOCATIONS:
Overall Officials: Alison Fox-Robichaud, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Holton D, Paton S, Conly J, Embree J, Taylor G, Thompson W. Central venous catheter-associated bloodstream infections occurring in Canadian intensive care units: A six-month cohort study. Can J Infect Dis Med Microbiol. 2006 May;17(3):169-76. doi: 10.1155/2006/781735. PMID 18418495
- [Result] Ziegler MJ, Pellegrini DC, Safdar N. Attributable mortality of central line associated bloodstream infection: systematic review and meta-analysis. Infection. 2015 Feb;43(1):29-36. doi: 10.1007/s15010-014-0689-y. Epub 2014 Oct 21. PMID 25331552
- [Derived] Pook M, Zamir N, McDonald E, Fox-Robichaud A. Chlorhexidine (di)gluconate locking device for central line infection prevention in intensive care unit patients: a multi-unit, pilot randomized controlled trial. Br J Nurs. 2022 Jul 21;31(14):S36-S46. doi: 10.12968/bjon.2022.31.14.S36. PMID 35856588
- [Derived] Zamir N, Pook M, McDonald E, Fox-Robichaud AE. Chlorhexidine locking device for central line infection prevention in ICU patients: protocol for an open-label pilot and feasibility randomized controlled trial. Pilot Feasibility Stud. 2020 Feb 18;6:26. doi: 10.1186/s40814-020-0564-9. eCollection 2020. PMID 32099661